CLINICAL TRIAL: NCT03462277
Title: DNA Methylation and Hydroxymethylation Levels in Patients With Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, doctor, Chongqing Medical University
Other Study IDs: 2016-39
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Coronary Heart Disease
Keywords: methylation; hydroxymethylation; atherosclerosis; coronary heart disease
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — human blood samples, human aortic tissues
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Control group was defined as people with negative findings in coronary angiograms.
- Coronary Heart Disease group: CHD patients was defined as at least one lesion in a coronary artery or branches in coronary angiograms.

SUMMARY:
The purpose of this trial is to investigate the relationship between DNA methylation and hydroxymethylation and the expression of DNMTs, TET family gene and the degree of coronary heart disease.

DETAILED DESCRIPTION:
1. To determine the levels of DNA methylation and hydroxymethylation with coronary heart disease.
2. To investigate the relationship between DNA methylation and hydroxymethylation and the degree of coronary atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

Male and Female. Patients older than 65 years old who are willing to participate in the study. CHD patients was defined as at least one lesion in a coronary artery or branches in coronary angiograms. Control group was defined as people with negative findings in coronary angiograms.

Exclusion Criteria:

Patients with concurrent infection or any documented inflammatory illness, such as arthritis or connective tissue diseases, or any other malignancy. Patients with a history of cardiomyopathy. Pregnant women. Severe hepatic dysfunction or End-stage renal failure. Uncontrolled hypertension.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with Coronary Heart Disease and Patients without Coronary Heart Disease.
  All patients underwent carotid ultrasound and coronary angiograms.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
DNA Methylation and Hydroxymethylation Levels | 1 month
  Collection of blood samples and measuring the samples by PCR and ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University; Dan Jiang, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China